CLINICAL TRIAL: NCT00557258
Title: Prevalence of Restless Legs Syndrome in Patients With Unpleasant Sensations of the Legs
Brief Title: Cross-Sectional Study: Prevalence of Restless Legs Syndrome in Patients With Unpleasant Sensations of the Legs
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.652
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

SUMMARY:
The proposed study is a Cross-sectional epidemiological study, performed in 330 primary care practices in Germany. The study will be conducted on a fixed day in November 2007.

Primary care surgeries throughout Germany will be asked to take part. The study material will be delivered to the surgery by a member of sales-force who will also explain the study conduct to the physician/staff. Physicians who want to take part in the study will send a signed contract to BI. Physicians will be trained to diagnose RLS.

All patients attending the participating surgeries on a fixed day will be invited to participate in the study. The patients will be handed a questionnaire to fill out while waiting for their appointment. No patient-related data apart from gender and year of birth will be recorded on the questionnaire and it will be ensured that no re-identification of patients is possible. Therefore, no written informed consent will be obtained from the participants.

The patient questionnaire will consist of the following items:

A screening questionnaire for RLS (according to Stiasny-Kolster et. al., data on file) Additional questions concerning the impact of the patients leg problems on daily life.

The practice staff will then collect the questionnaire. All patients who have answered question 1 (asking for unpleasant sensations of the legs) with ¿Yes¿ will subsequently be assessed for the diagnosis by the physician.

The physician fills out a second questionnaire, covering the following items:

Diagnosis (cause of leg problems) Concomitant diagnoses and therapies If the diagnosis of RLS was made: consequences (therapy)? Was the diagnosis of RLS pre-known? All completed questionnaires will be sent to data management by the surgery within 2 working days.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending one of the participating primary care surgeries on a fixed day
* Male or female patients of any age

Exclusion Criteria:

* Patients who only attend the practice to get a prescription and are not seen by the doctor on that day.
* Patients who are not able to understand the questionnaire due to mental impairment or language problems.
* Children and adolescents under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14956 (Actual)
Dates: Start 2007-11; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (251):
- Germany (251):
  - Boehringer Ingelheim Investigational Site, Aachen
  - Boehringer Ingelheim Investigational Site, Aalen
  - Boehringer Ingelheim Investigational Site, Ahlen
  - Boehringer Ingelheim Investigational Site, Altena
  - Boehringer Ingelheim Investigational Site, Altensteig
  - Boehringer Ingelheim Investigational Site, Altomünster
  - Boehringer Ingelheim Investigational Site, Alveslohe
  - Boehringer Ingelheim Investigational Site, Annaberg-Buchholz
  - Boehringer Ingelheim Investigational Site, Apolda
  - Boehringer Ingelheim Investigational Site, Artern
  - Boehringer Ingelheim Investigational Site, Aschersleben
  - Boehringer Ingelheim Investigational Site, Aub
  - Boehringer Ingelheim Investigational Site, Babenhausen
  - Boehringer Ingelheim Investigational Site, Bad Bevensen
  - Boehringer Ingelheim Investigational Site, Bad Buchau
  - Boehringer Ingelheim Investigational Site, Bad Essen
  - Boehringer Ingelheim Investigational Site, Bad Krozingen
  - Boehringer Ingelheim Investigational Site, Bad Laasphe
  - Boehringer Ingelheim Investigational Site, Bad Langensalza
  - Boehringer Ingelheim Investigational Site, Bad Schussenried
  - Boehringer Ingelheim Investigational Site, Bautzen
  - Boehringer Ingelheim Investigational Site, Bergholz-Rehbrücke
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Bernburg
  - Boehringer Ingelheim Investigational Site, Bernsdorf
  - Boehringer Ingelheim Investigational Site, Bevern
  - Boehringer Ingelheim Investigational Site, Biberach
  - Boehringer Ingelheim Investigational Site, Bienenbüttel
  - Boehringer Ingelheim Investigational Site, Birkenwerder
  - Boehringer Ingelheim Investigational Site, Bisingen
  - Boehringer Ingelheim Investigational Site, Bodelshausen
  - Boehringer Ingelheim Investigational Site, Bodenwöhr
  - Boehringer Ingelheim Investigational Site, Bornheim
  - Boehringer Ingelheim Investigational Site, Braunschweig
  - Boehringer Ingelheim Investigational Site, Bremen
  - Boehringer Ingelheim Investigational Site, Buckenhof
  - Boehringer Ingelheim Investigational Site, Buedelsdorf
  - Boehringer Ingelheim Investigational Site, Burgdorf, Hanover
  - Boehringer Ingelheim Investigational Site, Burgheim
  - Boehringer Ingelheim Investigational Site, Burgoberbach
  - Boehringer Ingelheim Investigational Site, Bückeburg
  - Boehringer Ingelheim Investigational Site, Bünde
  - Boehringer Ingelheim Investigational Site, Calbe
  - Boehringer Ingelheim Investigational Site, Calw
  - Boehringer Ingelheim Investigational Site, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site, Celle
  - Boehringer Ingelheim Investigational Site, Chemnitz
  - Boehringer Ingelheim Investigational Site, Cologne
  - Boehringer Ingelheim Investigational Site, Coppenbrügge
  - Boehringer Ingelheim Investigational Site, Cottbus
  - Boehringer Ingelheim Investigational Site, Cuxhaven
  - Boehringer Ingelheim Investigational Site, Daun
  - Boehringer Ingelheim Investigational Site, Dänischenhagen
  - Boehringer Ingelheim Investigational Site, Delligsen
  - Boehringer Ingelheim Investigational Site, Denkendorf
  - Boehringer Ingelheim Investigational Site, Dillingen
  - Boehringer Ingelheim Investigational Site, Donauwörth
  - Boehringer Ingelheim Investigational Site, Dormagen
  - Boehringer Ingelheim Investigational Site, Dorn-Dürkheim
  - Boehringer Ingelheim Investigational Site, Dortmund
  - Boehringer Ingelheim Investigational Site, Dörentrup
  - Boehringer Ingelheim Investigational Site, Dreieich
  - Boehringer Ingelheim Investigational Site, Dresden
  - Boehringer Ingelheim Investigational Site, Duisburg
  - Boehringer Ingelheim Investigational Site, Düren
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Edenkoben
  - Boehringer Ingelheim Investigational Site, Eisingen
  - Boehringer Ingelheim Investigational Site, Elsenfeld
  - Boehringer Ingelheim Investigational Site, Emsdetten
  - Boehringer Ingelheim Investigational Site, Eppelheim
  - Boehringer Ingelheim Investigational Site, Erftstadt
  - Boehringer Ingelheim Investigational Site, Erfurt
  - Boehringer Ingelheim Investigational Site, Erlangen
  - Boehringer Ingelheim Investigational Site, Erndtebrück
  - Boehringer Ingelheim Investigational Site, Eschau
  - Boehringer Ingelheim Investigational Site, Essen
  - Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site, Eutin
  - Boehringer Ingelheim Investigational Site, Extertal
  - Boehringer Ingelheim Investigational Site, Falkensee
  - Boehringer Ingelheim Investigational Site, Frankfurt
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site, Freising
  - Boehringer Ingelheim Investigational Site, Friedenfels
  - Boehringer Ingelheim Investigational Site, Friedrichsthal
  - Boehringer Ingelheim Investigational Site, Fulda
  - Boehringer Ingelheim Investigational Site, Fürstenwalde
  - Boehringer Ingelheim Investigational Site, Geiselhöring
  - Boehringer Ingelheim Investigational Site, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site, Gensingen
  - Boehringer Ingelheim Investigational Site, Germering
  - Boehringer Ingelheim Investigational Site, Gladbeck
  - Boehringer Ingelheim Investigational Site, Glashütten
  - Boehringer Ingelheim Investigational Site, Göttingen
  - Boehringer Ingelheim Investigational Site, Greiz
  - Boehringer Ingelheim Investigational Site, Großenkneten
  - Boehringer Ingelheim Investigational Site, Großenlüder
  - Boehringer Ingelheim Investigational Site, Grömitz
  - Boehringer Ingelheim Investigational Site, Haag
  - Boehringer Ingelheim Investigational Site, Hagen
  - Boehringer Ingelheim Investigational Site, Halle
  - Boehringer Ingelheim Investigational Site, Haltern
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Boehringer Ingelheim Investigational Site, Hamminkeln
  - Boehringer Ingelheim Investigational Site, Hanerau-Hademarschen
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Harsewinkel
  - Boehringer Ingelheim Investigational Site, Hartenstein
  - Boehringer Ingelheim Investigational Site, Hattorf
  - Boehringer Ingelheim Investigational Site, Heilbronn
  - Boehringer Ingelheim Investigational Site, Heinsberg
  - Boehringer Ingelheim Investigational Site, Herbertshofen
  - Boehringer Ingelheim Investigational Site, Herbrechtingen
  - Boehringer Ingelheim Investigational Site, Hermsdorf
  - Boehringer Ingelheim Investigational Site, Hohenhameln
  - Boehringer Ingelheim Investigational Site, Hosena
  - Boehringer Ingelheim Investigational Site, Hude
  - Boehringer Ingelheim Investigational Site, Ippesheim
  - Boehringer Ingelheim Investigational Site, Ispringen
  - Boehringer Ingelheim Investigational Site, Jahnsdorf
  - Boehringer Ingelheim Investigational Site, Jever
  - Boehringer Ingelheim Investigational Site, Jühnde
  - Boehringer Ingelheim Investigational Site, Jünkerath
  - Boehringer Ingelheim Investigational Site, Kahl am Main
  - Boehringer Ingelheim Investigational Site, Kalbach
  - Boehringer Ingelheim Investigational Site, Kamen
  - Boehringer Ingelheim Investigational Site, Kassel
  - Boehringer Ingelheim Investigational Site, Katzhütte
  - Boehringer Ingelheim Investigational Site, Kaufbeuren
  - Boehringer Ingelheim Investigational Site, Kirchardt
  - Boehringer Ingelheim Investigational Site, Kirchheim
  - Boehringer Ingelheim Investigational Site, Kirchlengern
  - Boehringer Ingelheim Investigational Site, Kitzingen
  - Boehringer Ingelheim Investigational Site, Kressbronn
  - Boehringer Ingelheim Investigational Site, Kronach
  - Boehringer Ingelheim Investigational Site, Kropp
  - Boehringer Ingelheim Investigational Site, Krumbach
  - Boehringer Ingelheim Investigational Site, Kuppenheim
  - Boehringer Ingelheim Investigational Site, Laatzen
  - Boehringer Ingelheim Investigational Site, Lahnau
  - Boehringer Ingelheim Investigational Site, Lahr
  - Boehringer Ingelheim Investigational Site, Lampertheim
  - Boehringer Ingelheim Investigational Site, Langen
  - Boehringer Ingelheim Investigational Site, Langenfeld
  - Boehringer Ingelheim Investigational Site, Lauf
  - Boehringer Ingelheim Investigational Site, Leer
  - Boehringer Ingelheim Investigational Site, Lehrberg
  - Boehringer Ingelheim Investigational Site, Leipzig
  - Boehringer Ingelheim Investigational Site, Lengefeld
  - Boehringer Ingelheim Investigational Site, Leonberg
  - Boehringer Ingelheim Investigational Site, Leverkusen
  - Boehringer Ingelheim Investigational Site, Lienen
  - Boehringer Ingelheim Investigational Site, Lohfelden
  - Boehringer Ingelheim Investigational Site, Lohra
  - Boehringer Ingelheim Investigational Site, Ludwigshafen
  - Boehringer Ingelheim Investigational Site, Lunzenau
  - Boehringer Ingelheim Investigational Site, Lüderitz
  - Boehringer Ingelheim Investigational Site, Lütjenburg
  - Boehringer Ingelheim Investigational Site, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mannheim
  - Boehringer Ingelheim Investigational Site, Marburg
  - Boehringer Ingelheim Investigational Site, Meerbusch
  - Boehringer Ingelheim Investigational Site, Meldorf
  - Boehringer Ingelheim Investigational Site, Mendig
  - Boehringer Ingelheim Investigational Site, Mengkofen
  - Boehringer Ingelheim Investigational Site, Meßstetten
  - Boehringer Ingelheim Investigational Site, Mindelheim
  - Boehringer Ingelheim Investigational Site, Mittweida
  - Boehringer Ingelheim Investigational Site, Moosburg
  - Boehringer Ingelheim Investigational Site, Mosbach
  - Boehringer Ingelheim Investigational Site, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, Mühlhausen
  - Boehringer Ingelheim Investigational Site, Mülheim
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Niederndodeleben
  - Boehringer Ingelheim Investigational Site, Nienburg
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Oberdorla
  - Boehringer Ingelheim Investigational Site, Oberursel
  - Boehringer Ingelheim Investigational Site, Oer-Erkenschwick
  - Boehringer Ingelheim Investigational Site, Olbernhau
  - Boehringer Ingelheim Investigational Site, Olfen
  - Boehringer Ingelheim Investigational Site, Osnabrück
  - Boehringer Ingelheim Investigational Site, Ostrach
  - Boehringer Ingelheim Investigational Site, Parey
  - Boehringer Ingelheim Investigational Site, Petershagen
  - Boehringer Ingelheim Investigational Site, Pirmasens
  - Boehringer Ingelheim Investigational Site, Plattling
  - Boehringer Ingelheim Investigational Site, Pleidelsheim
  - Boehringer Ingelheim Investigational Site, Potsdam
  - Boehringer Ingelheim Investigational Site, Pulheim
  - Boehringer Ingelheim Investigational Site, Rastede
  - Boehringer Ingelheim Investigational Site, Remscheid
  - Boehringer Ingelheim Investigational Site, Rhaunen
  - Boehringer Ingelheim Investigational Site, Roggendorf
  - Boehringer Ingelheim Investigational Site, Rossau
  - Boehringer Ingelheim Investigational Site, Rostock
  - Boehringer Ingelheim Investigational Site, Röthenbach
  - Boehringer Ingelheim Investigational Site, Saerbeck
  - Boehringer Ingelheim Investigational Site, Schorndorf
  - Boehringer Ingelheim Investigational Site, Schönau
  - Boehringer Ingelheim Investigational Site, Schönebeck
  - Boehringer Ingelheim Investigational Site, Schwarzenbach A Wald
  - Boehringer Ingelheim Investigational Site, Schwäbisch Gmünd
  - Boehringer Ingelheim Investigational Site, Schwerte
  - Boehringer Ingelheim Investigational Site, Seelow
  - Boehringer Ingelheim Investigational Site, Selfkant
  - Boehringer Ingelheim Investigational Site, Senftenberg
  - Boehringer Ingelheim Investigational Site, Siegen
  - Boehringer Ingelheim Investigational Site, Solingen
  - Boehringer Ingelheim Investigational Site, Sonsbeck
  - Boehringer Ingelheim Investigational Site, Sögel
  - Boehringer Ingelheim Investigational Site, Speyer
  - Boehringer Ingelheim Investigational Site, Sprendlingen
  - Boehringer Ingelheim Investigational Site, Stadland
  - Boehringer Ingelheim Investigational Site, Stadthagen
  - Boehringer Ingelheim Investigational Site, Straubing
  - Boehringer Ingelheim Investigational Site, Stuhr
  - Boehringer Ingelheim Investigational Site, Stutensee
  - Boehringer Ingelheim Investigational Site, Stuttgart
  - Boehringer Ingelheim Investigational Site, Suhl
  - Boehringer Ingelheim Investigational Site, Sulzbach
  - Boehringer Ingelheim Investigational Site, Sulzbach-Rosenberg
  - Boehringer Ingelheim Investigational Site, Teterow
  - Boehringer Ingelheim Investigational Site, Tettnang
  - Boehringer Ingelheim Investigational Site, Thaleischweiler-Fröschen
  - Boehringer Ingelheim Investigational Site, Troisdorf
  - Boehringer Ingelheim Investigational Site, Veilsdorf
  - Boehringer Ingelheim Investigational Site, Vellahn
  - Boehringer Ingelheim Investigational Site, Viernheim
  - Boehringer Ingelheim Investigational Site, Villingen-Schwenningen
  - Boehringer Ingelheim Investigational Site, Waghäusel
  - Boehringer Ingelheim Investigational Site, Wehrsdorf
  - Boehringer Ingelheim Investigational Site, Weibern
  - Boehringer Ingelheim Investigational Site, Weimar
  - Boehringer Ingelheim Investigational Site, Welzheim
  - Boehringer Ingelheim Investigational Site, Wemding
  - Boehringer Ingelheim Investigational Site, Wertingen
  - Boehringer Ingelheim Investigational Site, Wesel
  - Boehringer Ingelheim Investigational Site, Wesseling
  - Boehringer Ingelheim Investigational Site, Wetzendorf
  - Boehringer Ingelheim Investigational Site, Wetzlar
  - Boehringer Ingelheim Investigational Site, Wickede
  - Boehringer Ingelheim Investigational Site, Wiesbaden
  - Boehringer Ingelheim Investigational Site, Winsen
  - Boehringer Ingelheim Investigational Site, Wöbbelin
  - Boehringer Ingelheim Investigational Site, Zschocken
  - Boehringer Ingelheim Investigational Site, Zschopau
  - Boehringer Ingelheim Investigational Site, Zweibrücken
  - Boehringer Ingelheim Investigational Site, Zwickau